CLINICAL TRIAL: NCT04624685
Title: iStent Inject Trabecular Micro-Bypass System Continuation Post-Approval Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IG2M-104-CONT
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Long term follow up of subjects in the IDE study for iStent Inject to monitor safety

DETAILED DESCRIPTION:
To evaluate the long -term rate of clinically relevant complications associated with iStent inject® placement and stability in subjects who have completed participation of the IDE clinical trial (GC-008).

ELIGIBILITY:
Inclusion Criteria:

* Randomized subject followed for 24 months in the GC-008 study
* Able to understand study requirements
* Willing to attend scheduled follow-up exams for 5 years post-operatively
* Able and willing to provide written informed consent on the IRB approved Informed Consent Form

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 475 eyes of 475 subjects. This is based on the number of randomized subjects in the GC-008 study followed for 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
iStent inject Placement and Stability | 60 Months
  Rate of clinically relevant complications associated with iStent inject placement and stability.

SECONDARY OUTCOMES:
Sight-Threatening Adverse Events | 60 Months
  Rate of occurrence of sight-threatening adverse events

OTHER OUTCOMES:
Secondary Surgical Interventions | 60 Months
  Rate of Secondary Surgical Interventions
Adverse Events | 60 Months
  Rate of other adverse Events

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Arizona Advanced Eye Research Institute, Glendale, Arizona
  - Vold Vision, PLLC, Fayetteville, Arkansas
  - North Bath Eye Associates, Inc., Santa Rosa, California
  - Eye Center of northern Colorado, PC, Fort Collins, Colorado
  - Argus Research, Cape Coral, Florida
  - International Research Center, Tampa, Florida
  - Center for Sight, Venice, Florida
  - Clayton Eye Clinical Research, LLC., Morrow, Georgia
  - Chicago Eye Specialists, Chicago, Illinois
  - Arbor Center for Eye Care, Orland Park, Illinois
  - Stiles Eyecare Excellence, Overland Park, Kansas
  - D'Ambrosio Eye Care, Lancaster, Massachusetts
  - Kresge Eye Institute / Wayne State University, Detroit, Michigan
  - Discover Vision Centers, Independence, Missouri
  - Northern New Jersey Eye Institute, South Orange, New Jersey
  - Glaucoma Consultants of the Capital Region, Slingerlands, New York
  - Oklahoma eye Surgeons, PLLC, Oklahoma City, Oklahoma
  - Keystone Research, Austin, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - Parkhurst Nuvision, San Antonio, Texas
  - R and R Eye Resarch, LLC, San Antonio, Texas
  - Vistar Eye Center, Roanoke, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
  - The Eye Center of Racine and Kenosha, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: No